CLINICAL TRIAL: NCT02802956
Title: National Taiwan University Hospital, Taiwan
Brief Title: A Preliminary Feasibility Efficacy of Participation in Daily Life Promotion Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201509087RINC
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
Keywords: Life participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Daily Life Promotion Program
  Interventions: Other: Daily Life Promotion Program
- control group (Experimental): general rehabilitation treatment
  Interventions: Other: general rehabilitation treatment

INTERVENTIONS:
Other: Daily Life Promotion Program — Daily Life Promotion Program
  Arms: intervention group
Other: general rehabilitation treatment — general rehabilitation treatment
  Arms: control group

SUMMARY:
Efficacy of Participation in Daily Life Promotion Program for Patients with Chronic Stroke

DETAILED DESCRIPTION:
The purpose of this three-year research project is to develop an intervention program to promote participation in daily life for patients with chronic stroke and to evaluate its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stroke after 6 months.
* Must be able to follow orders and no other cognition impairment, Mini Mental State Examination scale must >20.

Exclusion Criteria:

* Clinical diagnosis of Dementia or Psychosis.
* Clinical diagnosis of Musculoskeletal disorders or Nervous system diseases.
* Patient with Congestive Heart Failure, Hypertension, Atrial fibrillation.
* Could not communication with others.
* Foreigner.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale(SIS) | one year
  quality of life measure

SECONDARY OUTCOMES:
Postural Assessment Scale for Stroke patients(PASS) | one year
  motor performance measure
Action Research Arm Test(ARAT) | one year
  motor performance measure
Fugl-Meyer Assessment(FMA) | one year
  motor performance measure
self-rated abilities for health practice scale | one year
  self-efficacy factors measure
WHO Quality of Life-BREF (Taiwan version) | one year
  quality of life measure
Taiwan Instrumental Activities of Daily Living(TIADL) | one year
  self-care ability measure
Barthel Index | one year
  self-care ability measure

CONTACTS AND LOCATIONS:
Overall Officials: I MING HSIAO, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: No